CLINICAL TRIAL: NCT07116057
Title: Phase I Clinical Trial of Autologous Folate Receptor-Alpha Redirected T Cells in Patients With FRa+ Cancers
Brief Title: MOv19-BBz CAR T Cells in FRa+ Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 858800 (UPCC #06525); R01CA260902 (NIH)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Non Small Cell Lung Cancer; Recurrent Lung Non-Small Cell Carcinoma
Keywords: NSCLC; CAR T cells; FRa+; lung cancer; lung adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung | interventions — CF regimen

STUDY DESIGN:
Intervention Model Description: Dose Level -1 (DL-1) will only be explored if ≥ 2 Treatment Limited Toxicities occur at any time in DL1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Dose Level 1 (DL1) (Experimental): single dose of 5x10(7) MOv19-BBz CAR T cells administered via intrapleural infusion following lymphodepleting chemotherapy
  Interventions: Biological: MOv19-BBz CAR T cells; Drug: Cyclophosphamide/Fludarabine; Device: FRa Expression Testing
- Dose Level -1 (DL-1) (Experimental): 2.5x10(7) MOv19-BBz CAR T cells adminstered via intrapleural infusion, following lymphodepleting chemotherapy. This dose level will only be explored if ≥ 2 TLTs occur at any time in DL1.
  Interventions: Biological: MOv19-BBz CAR T cells; Drug: Cyclophosphamide/Fludarabine; Device: FRa Expression Testing

INTERVENTIONS:
Biological: MOv19-BBz CAR T cells — Autologous T cells engineered to express an extracellular single chain variable fragment (scFv) with FRa specificity.
Drug: Cyclophosphamide/Fludarabine — Cytotoxic chemotherapy agents used for lymphodepletion prior to MOv19-BBz CAR T cell administration.
Device: FRa Expression Testing — Laboratory Developed Test used to determine subject eligibility

SUMMARY:
This is a Phase I open-label clinical trial to assess the safety, feasibility, and preliminary efficacy of intrapleural administration of MOv19-BBz CAR T cells in patients with FRa+ cancers. This study will be initiated in patients with metastatic or recurrent non-small cell lung cancer (NSCLC) only. Subjects will receive a single dose of MOv19-BBz CAR T cells via intrapleural infusion following lymphodepleting chemotherapy. Subjects without an existing intra-pleural catheter will have a temporary pleural catheter placed for the study. Subjects may initiate treatment with commercial checkpoint inhibitors per routine care beginning at least 28 days after receiving MOv19-BBz CAR T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Documentation of tumor FRa expression by IHC at the Hospital of the University of Pennsylvania (≥ 10% of tumor cells). Subjects must have archived tumor tissue available.
3. Disease-specific criteria:

   a. NSCLC Patients: i. Metastatic or recurrent lung adenocarcinoma with cytologically or pathologically confirmed malignant pleural effusion.

   ii. Failure of at least one prior line of standard of care therapy for advanced stage disease.
4. Patients must have evidence of active disease as defined by RECIST 1.1 criteria
5. Patients with asymptomatic CNS metastases that have been treated (and are off steroids for the treatment of CNS disease) are allowed. They must meet the following criteria

   1. No concurrent treatment for the CNS disease
   2. No progression of CNS metastasis on MRI at screening
   3. No evidence of leptomeningeal disease or cord compression
6. Adequate organ function deﬁned as:

   1. Serum creatinine ≤ 1.5 mg/dl or creatinine clearance ≥ 30 cc/min; Patient must not be on dialysis
   2. ALT/AST ≤ 3x upper limit of normal range
   3. Serum total bilirubin ≤ 1.5 mg/dl, unless the subject has Gilbert's syndrome (if so, serum total bilirubin must be ≤ 3.0 mg/dl)
   4. Must have a minimum level of pulmonary reserve deﬁned as < Grade 1 dyspnea and pulse oxygen > 92% on room air
   5. Left Ventricle Ejection Fraction (LVEF) ≥ 40% conﬁrmed by ECHO or MUGA
7. Male or female age ≥ 18 years
8. Eastern Cooperative Oncology Group (ECOG) Performance Status that is either 0 or 1
9. Subjects must be a possible clinical candidate for standard of care treatment with a commercial checkpoint inhibitor, as per physician-investigator assessment.

Exclusion Criteria:

1. Any clinically signiﬁcant pleural eﬀusion that cannot be drained with standard approaches.
2. Patients with signiﬁcant lung disease as follows:

   1. Patients with radiographic evidence of greater than lobar lymphangitic pulmonary involvement, greater than lobar bronchial wall thickening suggestive of peribronchial lymphatic disease extension, and/or evidence of extensive bilateral parenchymal metastatic burden.Note: "Greater than lobar" = "in more than 1 lobe".
   2. Patients with radiographic and/or clinical evidence of active radiation pneumonitis.
   3. Patients with radiographic evidence of underlying interstitial lung disease, including evidence of unresolved drug toxicity from any agent (e.g. chemotherapy, targeted agents, amiodarone, nitrofurantoin, etc.).
   4. Patients with radiographic evidence of signiﬁcant pleural effusion that is not readily amenable to minimally invasive drainage.
3. Active hepatitis B or hepatitis C infection
4. Any other active, uncontrolled infection
5. Class III/IV cardiovascular disability according to the New York Heart Association Classiﬁcation
6. Active invasive cancer, other than the proposed cancer included in this protocol, within 2 years prior to eligibility confirmation by a physician-investigator. [Note: non-invasive cancers treated with curative intent (e.g., non-melanoma skin cancer) may still be eligible].
7. Dependence on systemic steroids or immunosuppressant medications.
8. Pregnant or nursing (lactating) patients. Participants of reproductive potential must agree to use acceptable birth control methods
9. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10mg of prednisone daily. Patients with autoimmune neurologic diseases (such as MS) will be excluded.
10. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2040-10 (Estimated); Study Completion 2040-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events as assessed by CTCAE V5.0 | Up to 15 years post-MOv19-BBz CAR T cell administration
  Type, frequency, severity, and attribution of adverse events.
Occurrence of treatment-limiting toxicities (TLTs) | 28 days post-MOv19-BBz CAR T cell administration
  Unacceptable toxicity as defined by the protocol.

SECONDARY OUTCOMES:
Evaluate study feasibility | 6 months
  The proportion of enrolled subjects who are confirmed eligible and who receive study treatment as planned.
Objective Response Rate (ORR) | Up to 12 months following treatment with MOv19-BBz CAR T cells
  Proportion of subjects with confirmed CR or PR per RECIST 1.1 criteria.
Duration of Response (DOR) | Up to 15 years following treatment with MOv19-BBz CAR T cells
  Time from the date when confirmed CR or PR is first met, to the date of confirmed progressive disease, death due to any cause, or receipt of alternative anticancer therapy (excluding commercial immune checkpoint inhibitors as described by the study protocol); or it will be censored at the date of the last adequate assessment (whichever occurs first).
Progression Free Survival (PFS) | Up to 15 years following treatment with MOv19-BBz CAR T cells
  Duration from study treatment to disease progression, receipt of alternative anti-cancer therapy, or death.
Overall Survival (OS) | Up to 15 years following treatment with MOv19-BBz CAR T cell
  Duration of time from study treatment to the date of death, for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Haas, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No